CLINICAL TRIAL: NCT01186614
Title: Refractory Out-Of-Hospital Cardiac Arrest Treated With Mechanical CPR, Hypothermia, ECMO and Early Reperfusion
Acronym: CHEER
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: The Alfred (Other); Ambulance Victoria (Other Government)
Responsible Party: Principal Investigator, Ms. Rowan Frew, Director of Research and Ethics Unit, Bayside Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: project 160/10
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; ECMO; hypothermia; automated CPR; coronary intervention
MeSH Terms: conditions — Heart Arrest; Hypothermia | interventions — Hypothermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Novel treatment paradigm (Experimental): treatment protocol including - mechanical CPR, therapeutic hypothermia, ECMO, coronary intervention
  Interventions: Device: Automated CPR; Device: ECMO; Procedure: Coronary angiography; Procedure: Therapeutic Hypothermia

INTERVENTIONS:
Device: Automated CPR — Automated CPR utilised by paramedics to facilitate CPR during transport to hospital
  Other Names: Zoll Autopulse
Device: ECMO — Insertion of peripheral VA ECMO
Procedure: Coronary angiography — Coronary angiography and intervention where necessary will be performed following ECMO insertion
Procedure: Therapeutic Hypothermia — Paramedic initiated hypothermia with intravenous ice cold fluid and then continued for 24 hours (33 degrees)

SUMMARY:
Sudden out-of-hospital cardiac arrest (OHCA) is a leading cause of death in Australia. The most common cause of OHCA is a heart attack. The current treatment of OHCA is resuscitation by ambulance paramedics involving CPR, electrical shocks to the heart, and injections of adrenaline. In more than 50% of cases, paramedics are unable to start the heart and the patient is declared dead at the scene. Patients with OHCA who do not respond to paramedic resuscitation are not routinely transported to hospital because it is hazardous for paramedics to undertake rapid transport whilst administering chest compressions and there is currently no additional therapy available at the hospital that would assist in starting the heart.

However, a number of recent developments suggest that there may be a new approach to the resuscitation of this group of patients who would otherwise die.

Firstly, Ambulance Victoria have recently introduced portable battery powered machines that allow chest compressions to be safely and effectively delivered during emergency ambulance transport.

Second, The Alfred ICU will shortly be implementing a new protocol whereby the patient in cardiac arrest can immediately be placed on a heart-lung machine. This is known as extra-corporeal membrane oxygenation (ECMO).

Third, the brain can now be much better protected against damage due to lack of blood flow using therapeutic hypothermia which is the controlled lowering of body temperature from 37°C to 33°C. Clinical trials have demonstrated that this significantly decreases brain damage after OHCA.

Finally, The Alfred Cardiology service has an emergency service for reopening the blocked artery of the heart in patients who present with a sudden blockage of the heart arteries. This is currently not used in patients without a heart beat because of the technical difficulty of undertaking this procedure with chest compressions being undertaken.

This study proposes for the first time to implement all the above interventions when patients have failed standard resuscitation after OHCA. When standard resuscitation has proved futile, the patient will be transported to The Alfred with the mechanical chest compression device, cooled to 33°C, placed on ECMO, and then transported to the interventional cardiac catheter laboratory. The patient will then receive therapeutic hypothermia for 24 hours. Subsequent management will follow the standard treatment guidelines of The Alfred Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-59 years
* Out of hospital cardiac arrest due to presumed cardiac caus
* Chest compressions are commenced within 10 minutes by bystanders or emergency medical services
* Initial cardiac arrest rhythm of ventricular fibrillation
* Remains in cardiac arrest at the scene at 20 minutes after standard paramedic advanced cardiac life support (intubation, intravenous adrenaline)
* Autopulse machine is available
* Within 10 minutes ambulance transport time to The Alfred
* During normal working hours (9am-5pm, Monday to Friday)
* ECMO commences within 60 minutes of the initial collapse

Exclusion Criteria:

* Presumed non-cardiac cause of cardiac arrest such as trauma, hanging, drowning, intracranial bleeding
* Any pre-existing significant neurological disability
* Significant non-cardiac co-morbidities that cause limitations in activities of daily living such as COPD, cirrhosis of the liver, renal failure on dialysis, terminal illness due to malignancy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Survival to hospital discharge | At hospital discharge

SECONDARY OUTCOMES:
Neurologic recovery | At discharge
  Assessed by cerebral performance category
Time until ECMO insertion | On admission
neurologic biomarkers | Day 3
  neuron-specific enolase and S100β
Cardiac recovery | Days 1, 3, 5
  measured by echocardiography and cardiac biomakers including troponin, CK and BNP

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Bernard, MBBS MD, Principal Investigator — The Alfred
Locations (2):
- Australia (2):
  - Alfred Hospital, Melbourne, Victoria
  - Ambulance Victoria, Melbourne, Victoria